CLINICAL TRIAL: NCT06673290
Title: Different Doses of Sirolimus for the Treatment of Cystic Lymphatic Malformations
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, MD, PhD, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT20241029
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Lymphatic Malformation
Keywords: Lymphatic Malformation; sirolimus; Efficacy; Safety
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose of sirolimus (Experimental): The plasma trough concentration of sirolimus is maintained within the range of 5-8 ng/ml by adjusting sirolimus dose, for 1 year.
  Interventions: Drug: Sirolimus (RAPAMUNE)
- High dose of sirolimus (Active Comparator): The plasma trough concentration of sirolimus is maintained within the range of 10-15 ng/ml by adjusting sirolimus dose, for 1 year.
  Interventions: Drug: Sirolimus (RAPAMUNE)

INTERVENTIONS:
Drug: Sirolimus (RAPAMUNE) — Use of different doses of the same drug
  Other Names: Rapamycin; Rapamune

SUMMARY:
The purpose of this study is to compare the efficacy and safety of different concentration gradients of sirolimus in the treatment of cystic lymphatic malformation.

DETAILED DESCRIPTION:
Cystic lymphatic malformation is a disease caused by abnormal development of the lymphatic system, characterized by abnormal dilation and/or structural disorder of lymphatic vessels. These abnormalities may lead to accumulation of lymphatic fluid, causing local swelling, pain, and even affecting organ function. Cystic lymphatic malformation can occur anywhere in the body, including skin, soft tissue, internal organs, etc.

Sirolimus, also known as rapamycin, is an immunosuppressant mainly used to prevent rejection after organ transplantation. In recent years, studies have shown that sirolimus has certain potential in the treatment of lymphatic malformations.

However, long-term high-dose sirolimus treatment can cause some common complications, such as oral mucositis, which affects the quality of life of patients. More fine-grained control of rapamycin plasma concentrations may help improve the therapeutic effect and reduce the incidence of complications. Therefore, the investigators conducted this study to understand whether low-dose rapamycin is beneficial to the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a LM with the following characteristics:

  1. Male and female;
  2. Between 0 and 18 years of age;
  3. LM diagnosis was confirmed by local investigators and by consensus of our multidisciplinary vascular anomaly group at the West China Hospital of Sichuan University based on:

Biopsy; Compatible MRI findings; History and clinical features.

Exclusion Criteria:

1. Patients contraindicated for the administration of sirolimus (e.g., those with an allergy to sirolimus or other rapamycin analog)
2. Exposure to chemotherapy, embolization, corticosteroids, propranolol, sclerotherapy or any other investigational agents within 1 weeks before enrolment on study;
3. Patients had a history of a major surgery within 2 weeks before enrollment;
4. Patients who have a history of treatment with sirolimus or other mTOR inhibitor;
5. Any known evidence of significant local or systemic uncontrolled infection, defined as receiving intravenous antibiotics at the time of enrollment;
6. Concurrent severe and/or uncontrolled medical diseases that could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
7. Impairment of gastrointestinal function or chronic gastrointestinal disease that may significantly alter the absorption of sirolimus.
8. Patients with inadequate liver function:

   Total bilirubin higher than or equal to 1.5 × the upper limit of the normal (ULN) for age and alanine aminotransferase and aspartate aminotransferase higher than or equal to 2.5 × the ULN for age.
9. Patients with inadequate renal function:

   0-5 years of age maximum serum creatinine (mg/dL) of 0.8; 6-10 years of age maximum serum creatinine (mg/dL) of 1.0; 11-14 years of age maximum serum creatinine (mg/dL) of 1.2;
10. Adequate bone marrow function:

    Absolute neutrophil count lower than 1 × 109/L;
11. History of a malignancy within 5 years;
12. HIV infection or known immunodeficiency;
13. Indication for treatment with corticosteroids, vincristine, interferon-α, sirolimus, or tacrolimus for an indication other than IH;
14. Patients with an inability to participate in or follow-up during the study treatment and assessment plan;
15. Inability to give informed consent.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving an objective response at month 12 | 12 months
  Objective response was defined as ≥20% reduction in LM volume compared to that at baseline.

SECONDARY OUTCOMES:
The proportion of patients achieving an objective response at month 6 | 6 months
  Objective response was defined as ≥20% reduction in LM volume compared to that at baseline.
lesion responses | 6 and 12 months
  The primary endpoint was classified as follow: -Complete involution: 100% resolution of the measured LM; -Nearly complete involution was defined as decrease of ≥75% and <100%; -Partial involution was defined as decrease of ≥20% and <75%; -No change was defined as <20% increase and <20% decrease in the volumes of LM lesions; -Further growth was defined as ≥20% increase in the volume of index LM compared with the baseline volume measured. Lesion responses were overall lesion response rate and good lesion response rate. Overall lesion response comprised complete, nearly complete and partial involutions. Good lesion response comprised complete and nearly complete involutions.
Quality of life (QOL) in patients | 12 months
  Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Infant Scales (<2 years) or Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Scales (2-18 years) were used.
Disease sequelae | 12 months
  Disease sequelae were assessed by site investigators at month 12. The site investigators assessed patients' extremity swelling (if any), general physical activity and exercise levels.
Frequency of adverse events | 12 months
  Frequency of adverse events (e.g. gastrointestinal disorders, blood and lymphatic system disorders, metabolic disorders or other abnormal laboratory results, skin disorders and general disorders, etc.) collected by investigator and reported by parents. All adverse events were collected and graded according to Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0). The causality of the adverse event was determined by the multidisciplinary staff and was classified as definitively not related, probably not related, possibly related, probably related, or definitively related. Any dose reductions, interruptions, or cessations enacted at the discretion of the investigators were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghariani Fetoui N, Boussofara L, Gammoudi R, Belajouza C, Ghariani N, Denguezli M. Efficacy of sirolimus in the treatment of microcystic lymphatic malformation of the tongue. J Eur Acad Dermatol Venereol. 2019 Sep;33(9):e336-e337. doi: 10.1111/jdv.15628. Epub 2019 Apr 22. No abstract available. PMID 30980684
- [Background] Cai R, Yang X, Gu H, Chen H, Lin X. Comment on "Sirolimus for the treatment of verrucous venous malformation: A retrospective cohort study": Are we missing the lymphatic malformation component? J Am Acad Dermatol. 2023 Mar;88(3):e133-e134. doi: 10.1016/j.jaad.2018.08.050. Epub 2018 Sep 18. No abstract available. PMID 30240774
- [Background] Gu Y, Sebaratnam DF. Topical rapamycin and microcystic lymphatic malformations. J Am Acad Dermatol. 2024 Jan;90(1):e29-e30. doi: 10.1016/j.jaad.2023.06.066. Epub 2023 Sep 17. No abstract available. PMID 37717734
- [Background] Ozeki M, Endo S, Yasue S, Nozawa A, Asada R, Saito AM, Hashimoto H, Fujimura T, Yamada Y, Kuroda T, Ueno S, Watanabe S, Nosaka S, Miyasaka M, Umezawa A, Matsuoka K, Maekawa T, Hirakawa S, Furukawa T, Fumino S, Tajiri T, Takemoto J, Souzaki R, Kinoshita Y, Fujino A. Sirolimus treatment for intractable lymphatic anomalies: an open-label, single-arm, multicenter, prospective trial. Front Med (Lausanne). 2024 Feb 8;11:1335469. doi: 10.3389/fmed.2024.1335469. eCollection 2024. PMID 38390569
- [Background] Yonekura S, Komori T, Ishida Y, Kogame T, Kabashima K. Treatment With Topical Sirolimus for Recurrent Lymphatic Malformation of the External Urethral Meatus. JAMA Dermatol. 2022 Nov 1;158(11):1331-1332. doi: 10.1001/jamadermatol.2022.2793. PMID 36044195
- [Background] Strychowsky JE, Rahbar R, O'Hare MJ, Irace AL, Padua H, Trenor CC 3rd. Sirolimus as treatment for 19 patients with refractory cervicofacial lymphatic malformation. Laryngoscope. 2018 Jan;128(1):269-276. doi: 10.1002/lary.26780. Epub 2017 Aug 7. PMID 28782106
- [Background] Ozeki M, Fukao T. Generalized Lymphatic Anomaly and Gorham-Stout Disease: Overview and Recent Insights. Adv Wound Care (New Rochelle). 2019 Jun 1;8(6):230-245. doi: 10.1089/wound.2018.0850. Epub 2019 Jun 6. PMID 31236308
- [Background] Maruani A, Tavernier E, Boccara O, Mazereeuw-Hautier J, Leducq S, Bessis D, Guibaud L, Vabres P, Carmignac V, Mallet S, Barbarot S, Chiaverini C, Droitcourt C, Bursztejn AC, Lengelle C, Woillard JB, Herbreteau D, Le Touze A, Joly A, Leaute-Labreze C, Powell J, Bourgoin H, Gissot V, Giraudeau B, Morel B. Sirolimus (Rapamycin) for Slow-Flow Malformations in Children: The Observational-Phase Randomized Clinical PERFORMUS Trial. JAMA Dermatol. 2021 Nov 1;157(11):1289-1298. doi: 10.1001/jamadermatol.2021.3459. PMID 34524406